CLINICAL TRIAL: NCT01655615
Title: Co-venture: A Cluster Randomized Trial Investigating the Effects of Selective Intervention on Adolescent Cognitive Development and Addiction
Brief Title: Does Delaying Adolescent Substance Use Lead to Improved Cognitive Function and Reduce Risk for Addiction?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Justine's Hospital (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Patricia Conrod, Full Professor, St. Justine's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3427
Record Dates: First submitted 2012-03-14; First posted 2012-08-02 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Alcohol Related Disorders; Substance Related Disorders
Keywords: Adolescent cognitive development; mental disorders; Mood disorders; Alcohol-Related disorders; Mental disorders diagnosed in childhood; Substance related disorders
MeSH Terms: conditions — Alcohol-Related Disorders; Substance-Related Disorders; Mental Disorders; Mood Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Preventure programme (Experimental): The interventions are conducted using manuals which incorporate psycho-educational, motivational enhancement therapy and cognitive-behavioural (CBT) components, and include real life 'scenarios' shared by local youth in with similar personality profiles. In the first session, participants are guided in a goal-setting exercise, designed to enhance motivation to change behaviour. Psycho-educational strategies are then used to teach participants about the target personality variable and associated problematic coping behaviours like avoidance, interpersonal dependence, aggression, risky behaviours and substance misuse.
  Interventions: Behavioral: Preventure programme

INTERVENTIONS:
Behavioral: Preventure programme — The interventions are conducted using manuals which incorporate psycho-educational, motivational enhancement therapy and cognitive-behavioural (CBT) components, and include real life 'scenarios' shared by local youth in with similar personality profiles. In the first session, participants are guided in a goal-setting exercise, designed to enhance motivation to change behaviour. Psycho-educational strategies are then used to teach participants about the target personality variable and associated problematic coping behaviours like avoidance, interpersonal dependence, aggression, risky behaviours and substance misuse.

SUMMARY:
The Preventure Program is the first and only school-based alcohol and drug prevention program that has been shown to prevent onset and growth in alcohol and substance misuse in British and Canadian youth. Unlike universal programs that tend to promote generic coping skills and balance normative attitudes around substance use, this selected personality-targeted approach is based on a psychosocial model and validated by Dr Patricia Conrod and targets four personality-specific motivational pathways to substance misuse: Hopelessness, Anxiety Sensitivity, Impulsivity and Sensation Seeking, each associated with different motives for substance use, drug use profiles and patterns of non-addictive psychopathology.

As a primary goal of the Coventure project, the investigators propose a long-term trial of this intervention strategy to examine how this evidence-based intervention can reduce onset of substance use disorders in young people and related secondary mental health, academic and cognitive outcomes.

As a secondary goal, the investigators propose to use sensitive neuropsychological measures to examine how this evidence-based intervention can positively impact on cognitive development over the course of adolescence, to tease apart some of the mechanisms involved in the causal pathway from early onset substance use to poor cognitive development and long-term addiction outcomes.

DETAILED DESCRIPTION:
This is a cluster randomized design in which 31 high schools across Montreal, Canada will be randomly assigned to receive training and to deliver the program to two cohorts of Grade 7 students or to be trained and assisted in delivering the program to future Grade 7 cohorts. Assessment of participating students will occur annually from September to May until the end of high school year. Students will be assessed on personality, substance use, mental health and cognitive measures.

The program involves delivering specialized coping skills group workshops to students when they are in the 7th or 8th grade. About 45% of students in a given grade will be invited to participate in the workshops.

The workshops will focus on motivating children to understand how their personality style leads to certain emotional and behavioural reactions. They will be guided in learning cognitive behavioural skills on how to channel their strengths towards their long-term goals. Four different workshops will be run, focusing either on managing impulsivity, sensation seeking, anxiety sensitivity or negative thinking.

The students will first be asked to participate in a 45-60 minutes survey asking them about their personality, their strength and weaknesses, their risk-taking behaviour and their learning style.

Then, if their school has been trained to deliver the program, they might be invited to participate in two 90-minute workshops, delivered at school during class time or lunch hour. All children who agree to participate in the study will be invited to complete the same survey in each subsequent academic year for the next four years.

Primary outcomes:

1. Short-term: delayed onset of alcohol and substance use (up to two years post intervention)
2. Long-term: prevention of onset of substance use disorder (at 5th year follow-up).

Secondary intermediate outcomes are neuropsychological functions, for which two hypotheses will be investigated regarding the possible effects of delaying early substance use:

1. Global Effects Hypothesis: substance use and binge drinking will have global harmful effects on cognition and interventions that successfully prevent substance use onset will result in global improvements in cognitive function in participants who received the intervention relative to those randomized to control condition.
2. Critical Developmental Period Hypothesis: the toxic effects of alcohol and drug use are developmentally specific, so effects of interventions will be observed on cognitive processes that are maturing in adolescence, namely, executive functions and reward sensitivity, after controlling for general intelligence quotient (IQ) and memory function following procedure described by Séguin, et al (2004).

Secondary outcomes will be measures of poor mental health and functional cognitive measures such as academic achievement and school drop-out.

ELIGIBILITY:
Inclusion Criteria:

* Public or private high school
* Must have a Grade 7 cohort of at least 100 youth (up to 200), providing access to 45-90 high risk students per school Selection of high risk youth: Inclusion criteria for students are that they be enrolled in Grade 7 and that they have provided active assent and passive parental consent to participate in the longitudinal survey and randomised trial phases of this study. Participants who score 1 standard deviation above the school mean on one of four subscales of the Substance Use Risk Profile Scale will be selected to participate in the intervention groups, but all students will be followed on outcomes. There are no other exclusion criteria for participants.

Exclusion Criteria:

* Schools cannot be classified as having a majority of their students coded as special needs students, because these schools are smaller and the intervention protocol would have to be tailored for their particular needs

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2011-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Dep Ado: onset, frequency and binge items | Years 1, 2, 3,4 and 5
  The 'Detection of alcohol and drug problems in adolescents' questionnaire (DEP-ADO) is a self-report alcohol and illicit drug use measure in high-risk youth, including onset of drinking, binge drinking and illicit drug use. This tool has demonstrated good construct validity, internal consistency, test-retest and intermodal execution reliability in Quebec youth.

SECONDARY OUTCOMES:
Global cognitive function | Years 1, 2, 3,4 and 5
  1. A computerised adaptation of the Cultures Figure Task (CFT) is used to measure fluid intelligence. This task is based on two of the sections from Cattell's Culture Fair Intelligence Test: the linear pattern completion and matrix reasoning.
  ii. A computerised task based on the 'Dot Location' test, a subtest of the Child Memory Scales (CMS) is used to assess spatial memory. In this task, eight dots of the same colour are presented on a grid.
Executive function | Years 1, 2, 3,4 and 5
  Two tasks are used to assess executive functioning. i. 'Find the phone' is a spatial working memory task based on the Self-Order Pointing Task and is similar to the spatial working memory task of the Cambridge Neuropsychological Test Automated Battery (CANTAB).
  ii. An adaptation of the Go/No-Go Passive Avoidance Learning Paradigm (PALP) is used to assess cognitive control and response inhibition.
Functional cognitive measures | Years 1, 2, 3,4 and 5
  Data regarding academic achievement and school drop-out will be collected from the school administration.
Mental disorder symptoms | Years 1, 2, 3,4 and 5
  Depression and anxiety symptom severity over the past 12 months are measured using the Depression and Anxiety subscales from the Brief Symptoms Inventory. Conduct problems and hyperactivity/inattentive symptoms over the past 12 months are assessed according to the conduct and hyperactivity/inattentive subscales of the Strengths and Difficulties Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia J Conrod, PhD, Study Chair — Université de Montréal
Locations (1):
- CHU Sainte-Justine Research Center, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Lynch SJ, Stewart SH, Conrod P. Selective Personality-Targeted Intervention and the Escalation of Substance Use During Adolescence: A Secondary Analysis of A Cluster-Randomized Clinical Trial. JAMA Netw Open. 2025 Dec 1;8(12):e2550176. doi: 10.1001/jamanetworkopen.2025.50176. PMID 41632121
- [Derived] Wallace J, Boers E, Ouellet J, Conrod P. A Population-Based Analysis of the Temporal Association of Screen Time and Aggressive Behaviors in Adolescents. JAACAP Open. 2023 Aug 24;1(4):284-294. doi: 10.1016/j.jaacop.2023.08.002. eCollection 2023 Dec. PMID 39553451
- [Derived] Boers E, Afzali MH, Conrod P. A longitudinal study on the relationship between screen time and adolescent alcohol use: The mediating role of social norms. Prev Med. 2020 Mar;132:105992. doi: 10.1016/j.ypmed.2020.105992. Epub 2020 Jan 15. PMID 31954144
- [Derived] O'Leary-Barrett M, Pihl RO, Conrod PJ. Process variables predicting changes in adolescent alcohol consumption and mental health symptoms following personality-targeted interventions. Addict Behav. 2017 Dec;75:47-58. doi: 10.1016/j.addbeh.2017.06.022. Epub 2017 Jul 4. PMID 28692954